CLINICAL TRIAL: NCT03632681
Title: Interactions Between Metabolic, Cognitive and Reward Processes in Appetite - Effects of Intranasal Administration of Insulin
Brief Title: Effect of Intranasal Insulin on Cognitive Processes and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Queen Elizabeth Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RG_17-102
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: Cognitive processes; Reward processes; fMRI; Insulin
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin (Active Comparator): In this arm a single-dose of (160 IU/1.6ml) intranasal insulin will be administrated
  Interventions: Drug: Intranasal Insulin
- Placebo (Placebo Comparator): In this arm a single-dose intranasal placebo will be administrated
  Interventions: Drug: Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal Insulin — Intranasal insulin
  Other Names: Insulin; Actrapid
  Arms: Insulin
Drug: Intranasal Placebo — Intranasal placebo manufactured to mimic smell of insulin
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study investigates the effect of intranasal insulin on cognitive processes (behavioural and neural) in healthy lean and obese female adults. All subjects will receive a single-dose of intranasal insulin and/or placebo (on different days) before participating in several cognitive tasks.

DETAILED DESCRIPTION:
It is well established that eating behaviour is affected by metabolic signals (e.g. insulin, ghrelin, serotonin) and is also modulated via food reward processes. However, in humans, eating behaviour is a complex process, which involves habits, long-term goals and social interaction. Thus, recently it has been proposed that higher cognitive processes such as inhibitory control, attention and memory also modulate eating.

Insulin seems to be involved in both metabolic processes and cognitive processes. In the last decade it has been shown that intranasal administration of insulin decreases food intake, especially in women, and enhances thermogenesis and memory. In addition intranasal insulin administration has been shown to affect brain areas related to homeostatic control, reward and memory.

In the proposed study the investigators will examine the effect of intranasal insulin administration on eating, and on metabolic, reward and cognitive processes and their potential interplay. The investigators will also study the effect of body weight on the actions of insulin on these processes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* Age 18-65 years at start of the study
* Body Mass Index (BMI) between 18 and 25 kg/m2 for the lean group and between 30 and 40 kg/m2 for the obese group
* Right-handedness (including left-handers could bias the results because of the laterality of brain functions)
* Ability to give informed consent
* Fluent English speaking
* Willingness to be informed about chance findings of pathology

Exclusion Criteria:

* Subjects who have a non-removable metal object in or at their body, such as, for example: Heart pace-maker, artificial heart valve, metal prosthesis, implants or splinters, non-removable dental braces
* Tattoos, that are older than 15 years
* Claustrophobia
* Limited temperature perception and/or increased sensitivity to warming of the body
* Pathological hearing ability or an increased sensitivity to loud noises
* Lack of ability to give informed consent
* Operation less than three months ago
* Simultaneous participation in other studies that involve drugs intake or blood spending
* Acute illness or infection during the last 4 weeks
* Cardiovascular disorders (e.g., hypertrophic cardiomyopathy, long QT syndrome)
* Moderate or severe head injury
* Eating disorders
* No metabolic (e.g. metabolic disorder, diabetes, insulin resistance), psychological (e.g. depression) or neurological (e.g. epilepsy, headache disorder, multiple sclerosis, traumatic brain injuries) diseases or medication in relation to these diseases.
* Intake of any medication that can interfere with the drug or measurements.
* Current weight loss regimens, or more then 5kg weight loss in the last 3 months
* Smoking
* Current pregnancy or breastfeeding
* Current or past history of drug or alcohol dependency - alcohol consumption exceeding 12 units a week
* Food allergies (e.g. peanut allergy lactose and gluten intolerance) or vegetarian/vegan diet
* Disliking the study lunch

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation of gender identity
Enrollment: 64 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
fMRI brain response during inhibition to a food stimuli | 14 minutes
  Neural activation during correct inhibition food vs. non-food stimuli trail. Comparing the brain response when subjects correctly withhold for food vs a sports item.

SECONDARY OUTCOMES:
Delay discount of food reward | 5 minutes
  Area under the curve for delay of choosing a food item. Subjects have to choice between a certain amount of food now, or more (which varies between 1-20 pieces) food later (which will vary from 1 hour to 1 year).
Delay discount of money reward | 5 minutes
  Area under the curve for delay of choosing a amount of money. Subjects have to choice between a certain amount of money now, or more (which varies between 1-100 pound) money later (which will vary from 1 day, 1 months and 1 year).
fMRI brain activity in food picture task | 18 minutes
  Brain responses for food stimuli compared to non-food stimuli. The researchers will measure this by showing subjects food and non-food images while preforming and fMRI-scan and subtract activity during non-food images from the activity pattern when looking at food images.
Recall pictures | 5 minutes
  Recall accuracy. The researchers will count the correct amount of pictures remembered in this task and calculate % of pictures remembered in total, and differentiate between the three categories (high caloric/low caloric/control)
Recall words | 10 minutes
  Recall words. The researcher will count the correct amount of words remembered in this task
Emotional categorisation | 10 minutes
  Accuracy of category and reaction time will be measured for dislike or like words
Emotional recall part 1 | 4 minutes
  Recall words of liked and disliked words will be recorded in ECAT
Emotional recall part 1 | 10 minutes
  Accuracy of previous exposed or not exposed words will be measured
Cookie intake | 10 minutes
  Amount (kcal and gram) of cookies eaten will be measured
fMRI neural network during inhibition to a food stimuli | 14 minutes
  Functional connectivity during correct inhibition food vs. non-food stimuli trail.
fMRI brain responses during inhibition | 14 minutes
  Neural activation correct No-Go vs. Go trail. Subjects neural activation when they are instructed to go (press) when seeing toiletry or stationary items and react correctly compared to when subjects are instructed not to go (no press) when seeing a food or sport and withhold correctly

CONTACTS AND LOCATIONS:
Overall Officials: Maartje SPetter, PhD, Principal Investigator — Univerisity of Birmingham
Locations (1):
- Univerisity of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and data will be shared on Open Science Forum
Supporting Information: Study Protocol, ICF
Time Frame: The study protocol will be shared before including the first participant. The data will become available after the last participant has finished the study.
Access Criteria: All researchers
URL: https://osf.io